CLINICAL TRIAL: NCT01488539
Title: Implementation of an Evidence Based PTSD Treatment in Public Sector Settings
Brief Title: Implementation of an Evidence Based Post-Traumatic Stress Disorder (PTSD) Treatment in Public Sector Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: New York University (Other); Grady Health System (Other); Nathan Kline Institute for Psychiatric Research (Other); Georgetown University (Other); Harvard Medical School (HMS and HSDM) (Other); UConn Health (Other); VA New York Harbor Healthcare System (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Marylène Cloitre, Research Health Science Specialist, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLO0001AGG; 1R01MH086611-01A2 (NIH)
Record Dates: First submitted 2011-12-02; First posted 2011-12-08 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Stress Disorders, Post-Traumatic; PTSD; Adult Survivors of Child Abuse; Women; Interpersonal violence; psychological trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Trauma | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STAIR/NT (Experimental): Patients will receive STAIR/NT treatment
  Interventions: Behavioral: STAIR/NT treatment
- Treatment as Usual (TAU) (Other): Patients will receive Treatment as Usual (TAU)
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: STAIR/NT treatment — STAIR/NT is a two module, sequential treatment in which the first module emphasizes present-focused skills training in affective an interpersonal regulation (STAIR) for day-to-day life difficulties and the second module incorporates past-focused work on the processing of the trauma, using narrative therapy (NT). STAIR/NT is a cognitive behavioral treatment that can be flexibly applied allowing treatment tailored to the needs of the individual patient; may be as brief as 16 sessions and as long as 24.
  Arms: STAIR/NT
Behavioral: Treatment as Usual (TAU) — The Treatment as Usual intervention content varies from site to site and involve some combination of psychotherapy and pharmacotherapy. Treatment duration varies across sites and ranges from 30 to 45 sessions.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Researchers hope to learn whether a flexibly applied cognitive behavioral treatment for Post-Traumatic Stress Disorder (PTSD) is more effective than the psychotherapy usually provided in the clinic (called Treatment as Usual or TAU). Primary Hypothesis: STAIR/NT will be superior to TAU in improving PTSD symptoms at 28, 36 and 48 weeks post-randomization

DETAILED DESCRIPTION:
PTSD among women is a particularly pernicious and chronic disorder associated with significant psychiatric comorbidity, high rates of suicidality, substance abuse, self-injury and multiple traumatization including repeated sexual assault and domestic violence. Public-sector mental health services are the disproportionate recipient of traumatized women with between 62% to 98% of treatment seeking women reporting a history of trauma and of those, up to 40% carry a diagnosis of PTSD with various comorbidities. Over 40 single-site randomized trials of cognitive-behavioral therapy for PTSD have been conducted. However, to date, there are only two large-sample randomized clinical trials which have evaluated the effectiveness of such treatments in the community and both of them concerned military populations. This application proposes to evaluate the effectiveness of an evidence-based PTSD treatment in the context of a collaborative partnership of four public mental health clinics serving diverse populations. The intervention is a two module, sequential treatment (STAIR/NT) in which the first module emphasizes present-focused skills training in affective and interpersonal regulation (STAIR) for day-to-day life difficulties and the second module incorporates past-focused work on the processing of the trauma, using narrative therapy (NT). This cognitive behavioral treatment was specifically designed to treat high risk, multiply traumatized women with chronic PTSD and has been demonstrated to provide significant and clinically substantial relief from PTSD as well as improvement in emotion management and interpersonal functioning.

The investigators will assess the effectiveness of STAIR/NT compared to Treatment as Usual (TAU) in the context of every day clinical care. The study is a randomized, controlled repeated measures intent-to-treat design to assess STAIR/NT as compared to TAU at post-treatment and three and six-month follow-up. Four sites (Western Ontario, Boston, New York and Atlanta), each situated within a large public sector mental health network, will enroll 88 treatment-seeking women with PTSD related to interpersonal violence yielding a total of 352 study participants. The primary outcome will be PTSD symptom severity. Secondary outcomes will be negative mood regulation self-efficacy, interpersonal problems and general level of psychiatric impairment (GAF scores). Exploratory aims include the examination of the relationship between variations in treatment implementation and treatment outcome as well as the influence of patient characteristics and other contextual (therapist and organization) variables likely to impact implementation. The investigators will also introduce web-based technology as a resource intended to strengthen clinical networks and maintain use of study materials after the trial has ended.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of PTSD according to DSM-IV criteria with a CAPS score no lower than 40 (cf Weathers, Keane, & Davidson, 2001)
* PTSD symptoms that are a result of interpersonal violence
* at least one clear trauma memory
* Current age between 18 and 65
* If obtaining other (medication or psychosocial) treatment, must have completed at least a 3 month course of the treatment

Exclusion Criteria:

* Substance dependence and severe substance abuse disorders, current psychotic symptoms, unmedicated mania or bipolar disorder
* prominent current suicidal or homicidal ideation (a plan or intent versus a wish) or a suicide attempt within the past three months
* self-injurious behaviors in the last three months requiring medical attention
* Cognitive impairment indicated by chart diagnoses or observable cognitive difficulties
* Current involvement in a violent relationship defined as more than casual contact (e.g. dating or living with an abusive partner)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Clinician Assessed PTSD Symptom Severity | Baseline, 28, 36, 48 weeks
  Clinician Adminstered PTSD Scale for DSM-5 (CAPS-5) includes 20 items rated on a 5 point scale from 0 to 4. Possible total scores range from 0 to 80, with higher scores indicating more severe PTSD.
PTSD Diagnosis | Baseline, 28, 36, 48 weeks
  Clinician Adminstered PTSD Scale for DSM-5 (CAPS-5) assess the presence of PTSD diagnosis following the requirements indicated by DSM-5. These include the presence of 5 symtpom clusters that include re-experiencing symptoms, avoidance symptoms, alterations in mood and cognitions and hyperarousal.

SECONDARY OUTCOMES:
Emotion Regulation Problems | Baseline, 12, 28, 36, 48 weeks
  The DERS is a 36 item self-report measure where items are scored from 0 to 4 indicating how frequently the problem occurs. Possible total scores can range from 0 to 144 with higher scores indicating more frequent problems.
Interpersonal problems | Baseline, 12, 28, 36, 48 weeks
  The Inventory of Interpersonal Problems-32 (IIP-32) is a 32 item measure where items are scored from 0 to 4. Possible total scores range from 0 to 128 with higher scores indicating more severe problems.
Psychosocial Functioning | Baseline, 28, 36, 48 weeks
  SF-3 includes 3 items from the SF-36 which assess the impact of emotional problems on daily functioning

CONTACTS AND LOCATIONS:
Overall Officials: Marylene Cloitre, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (5):
- United States (5):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - Grady Health System, Atlanta, Georgia
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - New York University- Bellevue, New York, New York

REFERENCES:
- [Background] Cloitre M, Henn-Haase C, Herman JL, Jackson C, Kaslow N, Klein C, Mendelsohn M, Petkova E. A multi-site single-blind clinical study to compare the effects of STAIR Narrative Therapy to treatment as usual among women with PTSD in public sector mental health settings: study protocol for a randomized controlled trial. Trials. 2014 May 29;15:197. doi: 10.1186/1745-6215-15-197. PMID 24886235